CLINICAL TRIAL: NCT04551066
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of the Combination of PI3Kδ Inhibitor Parsaclisib and Ruxolitinib in Participants With Myelofibrosis
Brief Title: To Evaluate the Efficacy and Safety of Parsaclisib and Ruxolitinib in Participants With Myelofibrosis (LIMBER-313)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to futility.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 50465-313/LIMBER-313; 2020-003130-21 (EudraCT Number); NCT04816578 (obsolete NCT alias)
Record Dates: First submitted 2020-09-11; First posted 2020-09-16 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-09

CONDITIONS: Myelofibrosis; Primary Myelofibrosis; Post Essential Thrombocythemia Myelofibrosis; Post Polycythemia Vera Myelofibrosis
Keywords: INCB050465; ruxolitinib; parsaclisib; LIMBER; MF; Myelofibrosis; Myeloproliferative Neoplasms; Myoproliferative Neoplasms
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders | interventions — parsaclisib; ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A : parsaclisib + ruxolitinib (Experimental): Participants will receive parsaclisib and ruxolitinib starting from Day 1 for the duration of study, ruxolitinib dose will be determined by baseline platelet count.
  Interventions: Drug: parsaclisib; Drug: ruxolitinib
- Group B : placebo + ruxolitinib (Placebo Comparator): Participants will receive placebo and ruxolitinib starting from Day 1 for the duration of study, ruxolitinib dose will be determined by baseline platelet count.
  Interventions: Drug: ruxolitinib; Drug: placebo

INTERVENTIONS:
Drug: parsaclisib — parsaclisib will be administered QD orally
  Other Names: INCB050465
  Arms: Group A : parsaclisib + ruxolitinib
Drug: ruxolitinib — ruxolitinib will be administered BID orally
  Other Names: Jakafi; Jakavi
Drug: placebo — placebo will be administered QD orally
  Arms: Group B : placebo + ruxolitinib

SUMMARY:
The purpose of the study is to compare the efficacy of parsaclisib when combined with ruxolitinb versus placebo combined with ruxolitinib in participants with myelofibrosis.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind study of the combination of the PI3Kδ inhibitor parsaclisib or matching placebo and the JAK1/2 inhibitor ruxolitinib in participants with PMF or secondary MF (PPV-MF or PET-MF) with DIPSS risk category of intermediate or high. Prospective participants must have not received prior MF therapy with a JAK inhibitor or a PI3K inhibitor. After participants have been determined to be eligible for the study and completed the baseline symptom diary assessment for 7 days, they will be randomized to 1 of 2 treatment groups, with stratification for platelet count (≥ 100 × 10^9/L vs 50 to < 100 × 10^9/L inclusive) and DIPSS risk category (high vs intermediate-2 vs intermediate-1).

Once all enrolled participants completed the week 24 assessments the study will be unblinded and and participants randomized to placebo will have the opportunity to cross over to begin receiving parsaclisib, together with continued ruxolitinib, as long as hematology parameters are adequate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PMF, PPV-MF, or PET-MF.
* DIPSS risk category of intermediate-1, intermediate-2, or high.
* Palpable spleen of ≥ 5 cm below the left costal margin on physical examination at the screening visit.
* Active symptoms of MF at the screening visit, as demonstrated by the presence of a TSS of ≥ 10 using the Screening Symptom Form.
* Participants with an ECOG performance status score of 0, 1, or 2.
* Screening bone marrow biopsy specimen and pathology report(s) available that was obtained within the prior 2 months or willingness to undergo a bone marrow biopsy at screening/baseline; willingness to undergo bone marrow biopsy at Week 24 and every 24 weeks there after. Screening/baseline biopsy specimen must show diagnosis of MF.
* Life expectancy of at least 24 weeks.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Prior use of any JAK inhibitor.
* Prior therapy with any drug that inhibits PI3K (examples of drugs targeting this pathway include but are not limited to INCB040093, idelalisib, duvelisib, buparlisib, copanlisib, and umbralisib).
* Use of experimental drug therapy for MF or any other standard drug (eg, danazol, hydroxyurea) used for MF within 3 months of starting study drug and/or lack of recovery from all toxicities from previous therapy to ≤ Grade 1.
* Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications.
* Recent history of inadequate bone marrow reserve.
* Inadequate liver and renal function at screening.
* Active bacterial, fungal, parasitic, or viral infection that requires therapy.
* Active HBV or HCV infection that requires treatment or at risk for HBV reactivation.
* Known HIV infection.
* Uncontrolled, severe, or unstable cardiac disease that in the investigator's opinion may jeopardize the safety of the participant or compliance with the Protocol.
* Active invasive malignancy over the previous 2 years.
* Splenic irradiation within 6 months before receiving the first dose of study drug.
* Concurrent use of any prohibited medications.
* Active alcohol or drug addiction that would interfere with the ability to comply with the study requirements.
* Use of any potent CYP3A4 inhibitors or inducers within 14 days or 5 half lives(whichever is longer) before the first dose of study drug or anticipated during the study.
* Inadequate recovery from toxicity and/or complications from a major surgery before starting therapy.
* Currently breastfeeding or pregnant.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* History of Grade 3 or 4 irAEs from prior immunotherapy.
* Receipt of any live vaccine within 30 days of the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2024-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Assad, M.D, Study Director — Incyte Corporation
Locations (177):
- United States (36):
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - Mayo Clinic Rochester, Phoenix, Arizona
  - Sutter Health Alta Bates Summit Medical Center Absmc Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - CCARE, Fresno, California
  - California Research Institute (Cri), Los Angeles, California
  - UCLA School of Medicine, Los Angeles, California
  - Scripps Clinic, San Diego, California
  - Coastal Integrated Cancer Care-Cicc, San Luis Obispo, California
  - Stamford Hospital-Medical Oncology Hematology, Stamford, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - University of Kansas Hospital Authority, Westwood, Kansas
  - University of Kentucky-Markey Cancer Center, Lexington, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Midamerica Cancer Care, Kansas City, Missouri
  - New Jersey Hematology Oncology Associates Llc, Brick, New Jersey
  - Morristown Medical Center-Atlantic Health System, Morristown, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Westchester Medical Center Advanced Oncology and Infusion Center, Hawthorne, New York
  - Mount Sinai School of Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke Cancer Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Kaiser Permanente-Northwest, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Texas Oncology-Baylor Sammons Cancer Center, Dallas, Texas
  - Kelsey Seybold Clinic, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Renovatio Clinical, Spring, Texas
  - Providence Regional Medical Center Everett, Everett, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
- Austria (4):
  - Ordensklinikum Linz Gmbh Elisabethinen, Linz
  - Universitaetsklinikum St. Poelten, Saint Pï¿½LTEN
  - Hanusch-Krankenhaus Der Wiener Gebietskrankenkasse, Vienna
  - Hanusch-Krankenhaus Wiener Gebietskrankenkasse, Vienna
- Belgium (5):
  - A.Z. St.-Jan A.V., Bruges
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Grand Hospital de Charleroi, Charleroi
  - Jessa Ziekenhuis, Hasselt
  - AZ DELTA, Roeselare
- China (26):
  - Affiliated Hospital of Hebei University, Baoding
  - Peking University People'S Hospital (Pkuph) - Institute of Hematology, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangdong Provincial of People Hospital, Guangzhou
  - Nanfang Hospital, Guangzhou
  - The First Affiliated Hospital of Zhejiang University, Hangzhou
  - Harbin Institute of Hematology and Oncology, Harbin
  - Anhui Provincial Hospital, Hefei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Jinan Central Hospital, Jinan
  - The First Hospital of Lanzhou University, Lanzhou
  - Lanzhou University Second Hospital, Lanzhou
  - Jiangxi Provincial of People Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Zhongshan Hospital Fudan University, Shanghai
  - Shenzhen University Hospital, Shenzhen
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Provincial Peoples Hospital, Zhengzhou
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Odense University Hospital, Odense
- Helsinki University Central Hospital, Helsinki, Finland
- France (10):
  - Centre Hospitalier Universitaire Grenoble Alpes (Chu Grenoble Alpes) - Hopital Albert Michallon, La Tronche
  - Centre Hospitalier de Versailles - Hopital Andre Mignot, LE Chesnay-rocquencourt
  - Chu Limoges - Hopital Dupuytren, Limoges
  - Centre Hospitalier Universitaire de Nantes (Chu de Nantes) - Hotel-Dieu, Nantes
  - Chu Nimes, Nîmes
  - Ap-Hp Groupe Hospitalier Saint-Louis Lariboisiere Fernand-Widal Site Saint Louis (Paris), Paris
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hospital de La Miletrie, Poitiers
  - Chu de Rennes - Hospital Pontchaillou, Rennes
  - Centre Hospitalier de Roubaix, Roubaix
- Germany (4):
  - Universitatsklinikum Halle (Saale), Halle
  - Klinikum Kassel Gmbh, Kassel
  - Universitatsklinikum Magdeburg A.O.R., Magdeburg
  - Universitaetsmedizin Rostock, Rostock
- Israel (7):
  - Shamir Medical Center Formerly Assaf Harofeh Medical Center, BEER Yaaqov
  - Rambam Health Care Campus, Haifa
  - Hadassah Hebrew University Medical Center Ein Karem Hadassah, Jerusalem
  - Davidoff Cancer Center Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Ramat Hahayal, Tel Aviv
- Italy (19):
  - Lstituto Di Ematologia Lorenzo Ea.Seragnoli Universita Degli Studi Di Bologna - Policlinico S. Or, Bologna
  - Azienda Policlinico Vittorio Emanuele, Catania
  - Universita Degli Studi Di Genova - Facolta Di Medicina E Chirurgia, Genova
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori, Meldola
  - Istituto Di Ricovero E Cura A Carattere Scientifico (Irccs) Ospedale San Raffaele, Milan
  - Fondazione Irccs Ca Granda Ospedale Maggiore, Milan
  - Universita Di Napoli Federico Ii, Napoli
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Aormn Hospital Hematology and Bmt Center, Pesaro
  - Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli, Reggio Calabria
  - Universita Di Roma Tor Vergata, Roma
  - Universita Di Roma, Roma
  - Policlinico Universitario Agostino Gemelli Universita Cattolica Del Sacro Cuore, Roma
  - Policlinico Universitario Agostino Gemelli Universita Cattolica Del Sacro Cuore, Rome
  - Aou San Giovanni Di Dio E Ruggi D'Aragona, Salerno
  - Azienda Ospedaliera San Giuseppe Moscati, Taranto
  - Azienda Sanitaria Universitaria Friuli Centrale Asu Fc, Udine
  - A.O. Universitaria Ospedale Di Circolo E Fondazione Macchi, Varese
  - Azienda Ospedaliera Universitaria Integrata Verona (Ospedale Borgo Roma), Verona
- Japan (21):
  - Chiba Cancer Center, Chiba
  - University of Yamanashi Hospital, Chūō
  - Kyushu University Hospital, Fukuoka
  - Japanese Red Cross Society Himeji Hospital, Himeji-shi
  - Kansai Medical University Hospital, Hirakata
  - Tokai University Hospital, Isehara
  - Kagoshima University Hospital, Kagoshima
  - Hospital of the University of Occupation and Environmental Health, Kitakyushu-shi
  - Kobe City Medical Center General Hospital, Kobe
  - Kumamoto Shinto General Hospital, Kumamoto
  - University of Miyazaki Hospital, Miyazaki
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya
  - Osaka Metropolitan University Hospital, Osaka
  - Ogaki Municipal Hospital, Ōgaki
  - Dokkyo Medical University Saitama Medical Center, Saitama
  - Hokuyukai Sapporo Hokuyu Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Juntendo University Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Mie University Hospital, Tsu
  - Yokohama Municipal Citizens Hospital, Yokohama
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Akershus University Hospital, Lï¿½RENSKOG
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny Im. Andrzeja Mielckiego, Katowice
  - Pratia Hematologia Katowice, Katowice
  - Sp Zoz Szpital Uniwersytecki, Krakow
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
  - Institute of Hematology and Transfusion Medicine, Warsaw
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - THE CATHOLIC UNIVERSITY OF KOREA SEOUL ST. MARYï¿½S HOSPITAL, Seoul
  - Wonju Severance Christian Hospital, Wŏnju
- Spain (17):
  - Hospital General Unviersitario de Alicante, Alicante
  - Ico Hospital Germans Trias I Pujol, Badalona
  - Hospital Del Mar, Barcelona
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Ico-Hospital Duran I Reynals, Barcelona
  - Institut Catala Doncologia Ico - Hospital Duran I Reynals Location, Barcelona
  - Ico Hospital Germans Trias I Pujol, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitario Virgen de La Arrixaca, El Palmar
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Fundacian Jimnez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitari I Politecnic La Fe, Valencia
  - Hospital Universitario Doctor Peset, Valencia
- Turkey (Türkiye) (7):
  - Baskent University Adana Hospital, Adana
  - Gazi University Hospital Gazi University Faculty of Medicine, Ankara
  - Istanbul Medipol Universitesi Ibagcilar Medipol Mega Universitesi Hastanesi, Istanbul
  - Baskent University Istanbul Hospital, Istanbul
  - Ege University Hospital, Izmir
  - Dokuz Eylul University, Izmir
  - Ondokuz Mayis University Medicine Faculty, Samsun
- United Kingdom (6):
  - United Lincolnshire Hospitals, Boston
  - Gloucestershire Royal Hospital, Gloucester
  - Barts Health Nhs Trust - St Bartholomews Hospital, London
  - University College London Hospitals Nhs Foundation Trust, London
  - Sheffield Teaching Hospitals Nhs Foundation Trust - Weston Park Hospital, Sheffield
  - University Hospital of North Midlands Nhs Trust, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Related Info — https://www.incyteclinicaltrials.com/limber/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 93 study sites in Austria, Belgium, China, Denmark, Finland, France, Germany, Israel, Italy, Japan, Norway, Poland, South Korea, Spain, Turkey, the United Kingdom, and the United States.
Groups:
- Parsaclisib Plus Ruxolitinib: Participants were randomized to receive parsaclisib plus ruxolitinib beginning on Day 1 and continued on this regimen as long as it was tolerated and the participants did not meet any discontinuation criteria. Participants with a Baseline platelet count ≥100 × 10^9/Liter received ruxolitinib 15 milligrams (mg) twice daily (BID). Participants with a Baseline platelet count of 50 to < 100 × 10^9/Liters inclusive received ruxolitinib 5 mg BID. Participants were also stratified according to the Dynamic International Prognostic Scoring System (DIPSS) risk category (high versus intermediate-2 versus intermediate-1). Participants received parsaclisib at a dose of 5 mg once daily (QD).
- Placebo Plus Ruxolitinib: Participants were randomized to receive placebo plus ruxolitinib beginning on Day 1 and continued on this regimen until they left the study. Participants with a Baseline platelet count ≥100 × 10^9/Liter received ruxolitinib 15 mg BID. Participants with a Baseline platelet count of 50 to < 100 × 10^9/Liters inclusive received ruxolitinib 5 mg BID. Participants were also stratified according to the DIPSS risk category (high versus intermediate-2 versus intermediate-1). Participants received matching placebo at a dose of 5 mg QD. After 24 weeks, participants randomized to receive placebo plus ruxolitinib could have switched to treatment with parsaclisib plus ruxolitinib per the regimen received during the first 24 weeks of the study. Treatment continued for as long as the regimen was tolerated and the participant did not meet any discontinuation criteria.
Period: Overall Study
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Started | 125 | 127
Completed | 0 | 0
Not Completed | 125 | 127
Not completed — Death | 5 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Sponsor Decision | 104 | 117
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Awaiting Rollover to Another Study to Receive Ruxolitinib | 2 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Concomitant Diagnosis of Mature Plasmacytoid Dendritic Cell Proliferation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib | Total
Number analyzed (Participants) | 125 | 127 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (10.34) | 63.3 (10.90) | 63.3 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 49 | 98
  Male | 76 | 78 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 103 | 110 | 213
  Unknown or Not Reported | 15 | 10 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 80 | 84 | 164
  Black or African American | 1 | 1 | 2
  Asian | 33 | 31 | 64
  Not Reported | 10 | 10 | 20
  Captured as "Not Hispanic, Latino or Spanish" in Database | 1 | 0 | 1
  Turkish | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving ≥35% Reduction in Spleen Volume From Baseline to Week 24 as Measured by Magnetic Resonance Imaging [MRI] (or Computed Tomography [CT] Scan in Applicable Participants)
Description: Participants had an MRI of the upper and lower abdomen and pelvis to determine the spleen volume. A CT scan was substituted for participants who were not candidates for MRI or when MRI was not readily available. Determination of spleen length below the left costal margin was measured by palpation, using a flexible ruler provided by the sponsor.
Time Frame: Baseline; Week 24
Population: Intent-to-Treat (ITT) Population: all randomized participants. Treatment groups were defined according to the treatment assignment at randomization regardless of the actual study drug the participant took during their participation. Participants who had both Baseline and Week 24 measurements, or discontinued treatment before 27APR2023, or reached Week 24 before 27APR2023 but were missing Week 24 assessments were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 89 | 92
percentage of participants | 52.8 | 46.7
Statistical Analysis 1: Comparison: Parsaclisib Plus Ruxolitinib vs Placebo Plus Ruxolitinib; Test type: Superiority; p = 0.4224, Cochran-Mantel-Haenszel — calculated from Cochran Mantel-Haenszel test stratified by Baseline platelet count ≥100 x 10^9/Liters versus 50 to <100 x 10^9/Liters inclusive; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.71 to 2.26]

2. Secondary Outcome: Percentage of Participants Who Had a ≥50% Reduction in Total Symptom Score (TSS) From Baseline to Week 24 as Measured by the Myelofibrosis Symptom Assessment Form v4.0 (MFSAF v4.0) Diary
Description: Symptoms of myelofibrosis were assessed using the MFSAF v4.0 diary. The MFSAF v4.0 is composed of 7 individual symptom scores (fatigue, night sweats, itchiness, abdominal discomfort, pain under left ribs, early satiety, bone pain), each collected daily using a 0- (no symptoms) to 10-point (worst imaginable symptoms) scale. The daily TSS (0 to 70) is the sum of the 7 individual symptom scores collected on the same day. Higher TSS indicate more severe symptoms. The TSS was missing if there were any missing individual scores. Observations with missing dates were excluded from the analysis. The Baseline/Week 24 total score was defined as the average of the daily total scores from the last 7 days before the first dose of parsaclisib, placebo, or ruxolitinib/the Week 24 visit. The Baseline/Week 24 total scores was missing if there were ≥4 missing out of the 7 daily total scores.
Time Frame: Baseline; Week 24
Population: ITT Population. Participants who had both Baseline and Week 24 measurements, or discontinued treatment before 27APR2023, or reached Week 24 before 27APR2023 but were missing Week 24 assessments were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 89 | 98
percentage of participants | 34.8 | 38.8
Statistical Analysis 1: Comparison: Parsaclisib Plus Ruxolitinib vs Placebo Plus Ruxolitinib; Test type: Superiority; p = 0.5728, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.46 to 1.53]

3. Secondary Outcome: Change in TSS From Baseline to Week 24 as Measured by the MFSAF v4.0 Diary
Description: Symptoms of myelofibrosis were assessed using the MFSAF v4.0 diary. The MFSAF v4.0 is composed of 7 individual symptom scores (fatigue, night sweats, itchiness, abdominal discomfort, pain under left ribs, early satiety, bone pain), each collected daily using a 0- (no symptoms) to 10-point (worst imaginable symptoms) scale. The daily TSS (0 to 70) is the sum of the 7 individual symptom scores collected on the same day. Higher TSS indicate more severe symptoms. The TSS was missing if there were any missing individual scores. Observations with missing dates were excluded from the analysis. The Baseline/Week 24 total score was defined as the average of the daily total scores from the last 7 days before the first dose of parsaclisib, placebo, or ruxolitinib/the Week 24 visit. The Baseline/Week 24 total scores was missing if there were ≥4 missing out of the 7 daily total scores. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 24
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 119 | 125
scores on a scale
  Baseline | 19.8 (14.29) | 19.6 (13.07)
  Change from Baseline at Week 24: number analyzed (Participants) | 75 | 89
  Change from Baseline at Week 24 | -6.6 (12.36) | -6.8 (10.74)

4. Secondary Outcome: Time to the First ≥50% Reduction in TSS as Measured by the MFSAF v4.0 Diary
Description: as for outcome 2
Time Frame: Baseline; up to Week 24
Population: ITT Population, including censored participants. Censored participants didn't have a response at any time up to the last assessment date. Participants who didn't have a >=50% reduction in TSS was censored at the time of the last assessment. Participants with a DIPSS risk level of Low Risk Level (0 prognostic points) were excluded from the analysis. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method with log-log transformation.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 125 | 127
days | 67.0 [27.0 to 131.0] | 69.0 [35.0 to 143.0]
Statistical Analysis 1: Comparison: Parsaclisib Plus Ruxolitinib vs Placebo Plus Ruxolitinib; Test type: Superiority; p = 0.9490, Log Rank — calculated from log-rank test stratified by Baseline platelet count ≥100 × 10^9/Liters versus 50 to <100 × 10^9/Liters inclusive

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval between the randomization date and the date of death due to any cause.
Time Frame: up to 749 days
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 125 | 127
days | NA [NA to NA] — Due to participants rolling over to another study (NCT02955940), the follow-up time was not long enough to estimate the median and the upper and lower limits of the confidence interval. | NA [NA to NA] — Due to participants rolling over to another study (NCT02955940), the follow-up time was not long enough to estimate the median and the upper and lower limits of the confidence interval.

6. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE could therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE is defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug until 30 to 35 days after the last dose of parsaclisib/matching placebo or ruxolitinib.
Time Frame: up to 960 days
Population: Safety Population: all participants who received at least 1 dose of parsaclisib, placebo, or ruxolitinib. Treatment groups for this population were determined according to the actual treatment the participant received regardless of assigned study drug treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 125 | 127
Participants | 117 | 119

7. Secondary Outcome: Number of Participants With Any Grade 3 or Higher TEAE
Description: An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. A TEAE is defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug until 30 to 35 days after the last dose of parsaclisib/matching placebo or ruxolitinib. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grades 1 through 5. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: moderate; minimal, local or noninvasive intervention indicated; limiting instrumental activities of daily living (ADL). Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4: life-threatening urgent intervention indicated. Grade 5: death related to AE.
Time Frame: up to 960 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 125 | 127
Participants | 75 | 75

8. Secondary Outcome: Time of Onset of a ≥35% Reduction in Spleen Volume
Description: The time to the first ≥35% reduction in spleen volume is defined as the time from randomization to the first time participants had ≥35% reduction in spleen volume.
Time Frame: up to 925 days
Population: ITT Population, including censored participants. Censored participants didn't have a response at any time up to the last assessment date. Participants who didn't have a >=35% reduction in spleen volume were censored at the time of the last assessment. Participants with a DIPSS risk level of Low Risk Level (0 prognostic points) were excluded from the analysis. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method with log-log transformation.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 125 | 127
days | 88.0 [86.0 to 99.0] | 92.0 [87.0 to 253.0]
Statistical Analysis 1: Comparison: Parsaclisib Plus Ruxolitinib vs Placebo Plus Ruxolitinib; Test type: Superiority; p = 0.1085, Log Rank — [p-value comment as in outcome 4, analysis 1]

9. Secondary Outcome: Duration of Maintenance of a ≥35% Reduction in Spleen Volume
Description: The duration of ≥35% reduction from Baseline in spleen volume was defined as the interval between the first spleen volume measurement that was a ≥35% reduction from Baseline and the date of the first measurement that was no longer a ≥35% reduction from Baseline.
Time Frame: up to 925 days
Population: ITT Population. Participants with DIPSS risk level being low risk level (0 prognostic points) have been excluded from the analysis. Only those participants with a ≥35% reduction in spleen volume who then had a loss of ≥35% reduction in spleen volume with a 25% increase from NADIR were analyzed. If the maintenance end date was not observed before the database cutoff, the duration was censored at the last assessment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
Number analyzed (Participants) | 73 | 61
days | 505.0 [339.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants lost a >=35% reduction in spleen volume at the time of rollover to another study (NCT02955940). | NA [337.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants lost a >=35% reduction in spleen volume at the time of rollover to another study (NCT02955940).
Statistical Analysis 1: Comparison: Parsaclisib Plus Ruxolitinib vs Placebo Plus Ruxolitinib; Test type: Superiority; p = 0.6127, Log Rank — [p-value comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: up to 960 days
Description: Treatment-emergent adverse events, defined as AEs either reported for the first time or the worsening of pre-existing events after the first dose of study drug until 30 to 35 days after the last dose of parsaclisib/matching placebo or ruxolitinib, have been reported for the Safety Population.
Arm/Group | Parsaclisib Plus Ruxolitinib | Placebo Plus Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 6/125 | 3/127
Serious Adverse Events (participants affected / at risk) | 26/125 | 18/127
Other Adverse Events (participants affected / at risk) | 109/125 | 109/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parsaclisib Plus Ruxolitinib (N=125) | Placebo Plus Ruxolitinib (N=127)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood fibrinogen decreased (Investigations) | 1 (3) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster meningomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Hypoparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Intracranial mass (Nervous system disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Myelitis transverse (Nervous system disorders) | 1 (1) | 0 (0)
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parsaclisib Plus Ruxolitinib (N=125) | Placebo Plus Ruxolitinib (N=127)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 7 (9)
Abdominal pain (Gastrointestinal disorders) | 8 (10) | 8 (9)
Alanine aminotransferase increased (Investigations) | 18 (29) | 11 (14)
Anaemia (Blood and lymphatic system disorders) | 57 (70) | 68 (94)
Aspartate aminotransferase increased (Investigations) | 22 (38) | 10 (12)
Asthenia (General disorders) | 11 (13) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (9)
Blood alkaline phosphatase increased (Investigations) | 11 (12) | 2 (2)
Blood creatinine increased (Investigations) | 11 (13) | 6 (6)
COVID-19 (Infections and infestations) | 26 (27) | 15 (16)
Constipation (Gastrointestinal disorders) | 8 (8) | 11 (11)
Contusion (Injury, poisoning and procedural complications) | 8 (9) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 10 (11)
Cytomegalovirus infection (Infections and infestations) | 9 (9) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 21 (28) | 21 (30)
Dizziness (Nervous system disorders) | 6 (6) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 5 (6)
Fatigue (General disorders) | 11 (13) | 12 (14)
Headache (Nervous system disorders) | 7 (7) | 11 (14)
Hypertension (Vascular disorders) | 8 (8) | 5 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (5) | 7 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (5) | 7 (8)
Nausea (Gastrointestinal disorders) | 6 (7) | 10 (13)
Neutropenia (Blood and lymphatic system disorders) | 11 (15) | 5 (6)
Neutrophil count decreased (Investigations) | 7 (14) | 7 (11)
Night sweats (Skin and subcutaneous tissue disorders) | 7 (8) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 8 (9)
Platelet count decreased (Investigations) | 29 (48) | 19 (38)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 9 (10)
Pyrexia (General disorders) | 9 (11) | 8 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 26 (31) | 21 (33)
Urinary tract infection (Infections and infestations) | 5 (5) | 7 (7)
Vomiting (Gastrointestinal disorders) | 8 (8) | 8 (10)
Weight increased (Investigations) | 7 (7) | 5 (7)
White blood cell count decreased (Investigations) | 8 (16) | 5 (5)

LIMITATIONS AND CAVEATS:
Due to participants rolling over to another study (NCT02955940), no participants randomized to receive placebo plus ruxolitinib switched to treatment with parsaclisib plus ruxolitinib.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT04551066/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT04551066/SAP_001.pdf